CLINICAL TRIAL: NCT00377026
Title: FirstWIND: Weight Loss Interventions After Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Wanda Nicholson, MD, MPH, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: M051633
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2009-06-19 (Estimated); Status verified 2009-06

CONDITIONS: Overweight; Obesity
Keywords: weight loss; postpartum; weight retention
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lifestyle (Experimental): participants receive lifestyle intervention
  Interventions: Behavioral: lifestyle intervention

INTERVENTIONS:
Behavioral: lifestyle intervention — Lifestyle modification including individual sessions with an interventionist to discuss dietary intake and exercise. Group sessions with other participants randomized to the lifestyle intervention to discuss lifestyle modification and group exercise.

SUMMARY:
This a pilot intervention study in which postpartum women will be randomized to receive a 6-month postpartum weight loss intervention or usual care.

DETAILED DESCRIPTION:
Overweight and obesity affect over 15 million adult women in the United States. Postpartum weight retention has been shown to be one factor contributing to weight retention, obesity and possible development of type 2 diabetes. African-American women and other minority women are at especially high risk for the development of obesity and type 2 diabetes. We propose to pilot a six-month postpartum-specific lifestyle intervention among urban-based, postpartum African-American women.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women with a pre-pregnancy or first trimester body mass index of 28 or greater or a history of gestational diabetes in the most recent pregnancy.

Exclusion Criteria:

* Current cardiac disease or serious chronic disease, including cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
weight loss | baseline, 3 months, and 6 months

SECONDARY OUTCOMES:
health status | baseline and six months
body mass index | baseline, 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wanda Nicholson, MD, MPH, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States